CLINICAL TRIAL: NCT00772590
Title: Randomised Double-blind Placebo Controlled Study to Measure the Effect of Antiretroviral Therapy (ART) Intensification With Raltegravir and/or Hyper-immune Bovine Colostrum on CD4+ T Cell Count in ART Treated, HIV-1 Infected Individuals With Suboptimal CD4+ T Cell Responses
Brief Title: Antiretroviral Therapy Intensification With Raltegravir or Addition of Hyper-immune Bovine Colostrum in HIV-1 Infected Patients With Suboptimal CD4+ T Cell Response
Acronym: CORAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kirby Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NCHECR-CORAL 1
Record Dates: First submitted 2008-10-14; First posted 2008-10-15 (Estimated); Results first posted 2012-08-24 (Estimated); Last update posted 2012-08-24 (Estimated); Status verified 2012-07

CONDITIONS: HIV Infections
Keywords: HIV; antiretroviral therapy intensification; suboptimal CD4+ T cell response; virological suppression; bovine colostrum; raltegravir
MeSH Terms: conditions — HIV Infections | interventions — Raltegravir Potassium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Raltegravir, bovine colostrum (Experimental): Raltegravir and hyper-immune bovine colostrum
  Interventions: Drug: raltegravir and hyper-immune bovine colostrum
- Hyper-immune bovine colostrum (Experimental): Hyper-immune bovine colostrum and Raltegravir placebo
  Interventions: Drug: Hyper-immune Bovine Colostrum
- Raltegravir (Experimental): Raltegravir and Hyper-immune Bovine Colostrum Placebo
  Interventions: Drug: Raltegravir
- Placebo (Placebo Comparator): Raltegravir placebo and hyper-immune bovine colostrum placebo
  Interventions: Other: raltegravir placebo; Other: Hyper-immune Bovine Colostrum placebo

INTERVENTIONS:
Drug: Raltegravir — Tablets, 400mg, twice daily
  Arms: Raltegravir
Drug: Hyper-immune Bovine Colostrum — Tablet, 1800mg, twice daily
  Arms: Hyper-immune bovine colostrum
Other: raltegravir placebo — One tablet, twice daily
  Other Names: placebo
  Arms: Placebo
Other: Hyper-immune Bovine Colostrum placebo — Three tablets twice daily
  Arms: Placebo
Drug: raltegravir and hyper-immune bovine colostrum — 400mg twice daily raltegravir and 1800mg twice daily of hyper-immune bovine colostrum
  Other Names: Raltegravir + hyper-immune bovine colostrum
  Arms: Raltegravir, bovine colostrum

SUMMARY:
A research study to measure the effect on CD4 counts of adding to current anti-retroviral regimen raltegravir with or without hyper-immune bovine colostrum.

DETAILED DESCRIPTION:
The primary objective of this study is to measure the effect on CD4+ T cell outcome as measured by the mean time weighted CD4+ T cell count change over 24 weeks of two interventions: (I) cART intensification with raltegravir and (II) cART combined with hyper-immune bovine colostrum in HIV-1 infected individuals who have failed to achieve a CD4+ T cell count greater than 350 cells/µL despite persistent HIV plasma viraemia below 50 copies/mL on cART.

Eligible patients will be randomised to one of four arms. I. Raltegravir + hyper-immune bovine colostrum placebo II. Raltegravir placebo + hyper-immune bovine colostrum III. Raltegravir + hyper-immune bovine colostrum IV. Raltegravir placebo + hyper-immune bovine colostrum placebo

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV-1 infection
* Age >18 years
* Signed informed consent
* Receiving combination ART (cART) for at least 12 months with a stable cART regimen for a minimum of 6 months. A formulation change or modification of dosage schedule is acceptable (for example ritonavir - boosted lopinavir capsules for tablets, abacavir (ABC) or tenofovir (TDF) and lamivudine (3TC) or emtricitabine (FTC) as single agents for ABC/3TC or TDF/FTC fixed dose combinations)
* Two consecutive plasma HIV RNA viral load measurements <50 (or <400 copies/mL depending upon lowest level of detection of the local assay) in the 9 months preceding the screening visit. A single isolated HIV RNA viral load >50 (or >400) copies/mL will not exclude the patient provided the viral load result >50 (or 400) copies/mL on therapy follows a previous result <50 (or 400) copies/mL, and there is a follow-up result <50 copies/mL at least one week following the >50 (or 400) copies/mL reading in the absence of a change to any component of the ART regimen.
* CD4+ T cell count <350 cells/µL throughout the 6 months preceding the screening visit with <50 cells/µL increase in the last 12 months

Exclusion Criteria:

* Receiving a cART regimen containing an integrase inhibitor
* Anticipated change of cART in the 24 weeks following randomisation
* Participating in study with an investigational compound or device within 30 days of signing informed consent
* Use of immune modulating therapies or immunosuppressive medications within 60 days prior to study entry. Patients using inhaled or nasal steroids are not excluded
* Pregnant or breastfeeding woman
* Cow's milk allergy
* Concurrent treatment with phenobarbitol, phenytoin or rifampicin.
* A known cause of impaired CD4+ T cell gain: for example, patients with splenomegaly or individuals whose current cART regimen contains both tenofovir and didanosine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2009-03; Primary Completion 2010-03 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sean Emery, BSc (Hons), PhD, Principal Investigator — National Centre in HIV Epidemiology and Clinical Research, University of New South Wales

REFERENCES:
- [Result] Byakwaga H, Kelly M, Purcell DF, French MA, Amin J, Lewin SR, Haskelberg H, Kelleher AD, Garsia R, Boyd MA, Cooper DA, Emery S; CORAL Study Group. Intensification of antiretroviral therapy with raltegravir or addition of hyperimmune bovine colostrum in HIV-infected patients with suboptimal CD4+ T-cell response: a randomized controlled trial. J Infect Dis. 2011 Nov 15;204(10):1532-40. doi: 10.1093/infdis/jir559. Epub 2011 Sep 19. PMID 21930607

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 100 patients were screening at 20 clinical sites in Australia
Pre-assignment Details: 25 of 100 patients screened did not meet study inclusion criteria and were excluded from study
Groups:
- Raltegravir + Hyper-immune Bovine Colostrum: Raltegravir and hyper-immune bovine colostrum
Period: Overall Study
Arm/Group | Raltegravir + Hyper-immune Bovine Colostrum | Hyper-immune Bovine Colostrum | Raltegravir | Placebo
Started | 19 | 19 | 18 | 17
Completed | 19 | 19 | 18 | 17
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Raltegravir + Hyper-immune Bovine Colostrum | Hyper-immune Bovine Colostrum | Raltegravir | Placebo | Total
Number analyzed (Participants) | 19 | 19 | 18 | 17 | 73
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 18 | 18 | 17 | 16 | 69
  >=65 years | 1 | 1 | 1 | 1 | 4
Age Continuous [Mean (Standard Deviation); unit: years] | 52 (11) | 56 (9) | 50 (10) | 55 (10) | 53 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 0 | 1 | 4
  Male | 17 | 18 | 18 | 16 | 69
Region of Enrollment [Number; unit: participants]
  Australia | 19 | 19 | 18 | 17 | 73

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline CD4+ Cell Count
Description: Comparison of normalised mean change from baseline CD4+ cell count
Time Frame: 24 weeks
Population: intention to treat (ITT) - all randomised patients who commenced randomly assigned therapy and who had at least one on-study visit.
Measure: Mean (Standard Deviation); unit: Cells/microlitre
Arm/Group | Raltegravir + Hyper-immune Bovine Colostrum | Hyper-immune Bovine Colostrum | Raltegravir | Placebo
Number analyzed (Participants) | 19 | 19 | 18 | 17
Cells/microlitre | 8.62 (32.19) | 2.68 (35.8) | 8.68 (44.58) | 21.87 (34.8)
Statistical Analysis 1: Comparison: Raltegravir + Hyper-immune Bovine Colostrum vs Hyper-immune Bovine Colostrum vs Raltegravir vs Placebo; Test type: Superiority or Other; p < 0.01, ANOVA

ADVERSE EVENTS:
Time Frame: Baseline to week 24
Arm/Group | Raltegravir + Hyper-immune Bovine Colostrum | Hyper-immune Bovine Colostrum | Raltegravir | Placebo
Serious Adverse Events (participants affected / at risk) | 1/19 | 0/19 | 1/18 | 1/17
Other Adverse Events (participants affected / at risk) | 0/19 | 0/19 | 0/18 | 0/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Raltegravir + Hyper-immune Bovine Colostrum (N=19) | Hyper-immune Bovine Colostrum (N=19) | Raltegravir (N=18) | Placebo (N=17)
Hosp. For cellulitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hosp. for possible Influenza A (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hosp. for chest pain (Cardiac disorders) | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Effect of interventions only measured in peripheral blood

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No